CLINICAL TRIAL: NCT05644340
Title: Feasibility and Safety Properties of Metabolic Flow Anesthesia Driven by Automated Gas Control in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associate Professor, Istanbul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2019/154
Record Dates: First submitted 2022-11-29; First posted 2022-12-09 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia
Keywords: pediatric anesthesia; metabolic flow anesthesia; low flow anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automated Gas Flow Group using speed 8 to reach targeted end-tidal sevoflurane concentration (Active Comparator): Pediatric patients who are operated under general anesthesia using automated gas flow which is set to speed 8 to achieve targeted end-expiratory sevoflurane concentration (MAC 1.2) will be included in the study. Automated gas flow provides a gas mixture in different proportions which is automatically generated and consists of sevoflurane, oxygen and air. Inspired and end-tidal concentrations of sevoflurane, oxygen and air will be available on the anesthesia ventilator screen which will be recorded accordingly in15-minute intervals.
  Interventions: Procedure: Speed 8 (Fast balancing gas flow)
- Automated Gas Flow Group using speed 4 to reach targeted sevoflurane concentration (Active Comparator): Pediatric patients who are operated under general anesthesia using automated gas flow which is set to speed 4 to achieve targeted end-expiratory sevoflurane concentration (MAC 1.2) will be included in the study. Automated gas flow provides a gas mixture in different proportions which is automatically generated and consists of sevoflurane, oxygen and air. Inspired and end-tidal concentrations of sevoflurane, oxygen and air will be available on the anesthesia ventilator screen which will be recorded accordingly in15-minute intervals.
  Interventions: Procedure: Speed 4 (Medium speed balancing gas flow)

INTERVENTIONS:
Procedure: Speed 8 (Fast balancing gas flow) — General anesthesia will be induced via intravenous agents, and anesthesia maintenance will be provided via inhalation for all the patients. The maintenance will be provided with sevoflurane using automated gas flow with the selected speed of 8. The anesthesia machine indicates amount of sevoflurane inhaled, inspired and exhaled oxygen, carbon dioxyde, air and sevoflurane concentrations. Accordingly these data and actual flow rate will be recorded every 15 minutes.
  Arms: Automated Gas Flow Group using speed 8 to reach targeted end-tidal sevoflurane concentration
Procedure: Speed 4 (Medium speed balancing gas flow) — General anesthesia will be induced via intravenous agents, and anesthesia maintenance will be provided via inhalation for all the patients. The maintenance will be provided with sevoflurane using automated gas flow with the selected speed of 4 (Medium speed). The anesthesia machine indicates amount of sevoflurane inhaled, inspired and exhaled oxygen, carbon dioxyde, air and sevoflurane concentrations. Accordingly these data and actual flow rate will be recorded every 15 minutes.
  Arms: Automated Gas Flow Group using speed 4 to reach targeted sevoflurane concentration

SUMMARY:
Low flow anesthesia was considered to be causing rebreathing, hypoxia and hypercarbia in the past. However, developing technologies made anesthesia ventilators safer. Low flow anesthesia is proved to be safe and cost-effective for almost a decade, and newer anesthetic machines with automated gas flow and metabolic flow anesthesia (<0.3 L/min gas flow) features are now becoming prominent.

The literature still lacks of pediatric data regarding the cost analysis and safety profile of low flow and especially in metabolic flow anesthesia. In this study, it is aimed to observe inhaled agent expenditure of automated gas flow anesthesia which reaches metabolic flow limits in pediatric patients. For that, automated gas flow will be set to provide a desired end-tidal sevoflurane concentration during general anesthesia. Accordingly, inspired fraction of oxygen and air values will be recorded in 15-minute intervals. Primary outcome will be the inhaled agent (sevoflurane) amount wasted in milliliters for both inhaled agent maintenance speed (8-fast and 4-slow). Secondarily, delta value of set and detected inspired fraction of oxygen (DeltaFiO2=DetectedFiO2-SetFiO2) will be analyzed. DeltaFiO2 higher than 5 units will be accepted as "unsafe" gas mixture, and the incidence will be evaluated. Secondary outcomes will also include duration of emergence from anesthesia including both extubation and obeying verbal commands.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric surgery patients
* Elective or Semielective surgeries
* Patients suitable for inhalation anesthesia

Exclusion Criteria:

* Emergency surgery
* Patients who are contraindicated for inhalation anesthesia

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Total amount of sevoflurane consumed | up to 3 hours
  At the end of the surgery, total amount of sevoflurane, which is indicated on the anesthesia machine screen, will be recorded in milliliters

SECONDARY OUTCOMES:
Time to extubation after inhalation anesthesia stop | Up to 45 minutes
  Time between the inhalation anesthesia stop and extubation in minutes
Time to cooperation after inhalation anesthesia stop | Up to 2 hours
  Time between the inhalation anesthesia stop and cooperation to verbal impulses in minutes
Delta Oxygen Concentration | up to 2 hours
  The adjusted oxygen fraction (generally 40%) minus the actual inhaled oxygen fraction will provide the delta value. The data will be recorded every 15-minute during the surgery, and delta >%5 will be considered as "unsafe"

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)